CLINICAL TRIAL: NCT04544696
Title: Pharmacists in Detecting Opioid Misuse Using the Prescription Opioid Misuse Index (POMI): Survey in a Region in the South of France, Occitanie-Est
Brief Title: Pharmacist for Detecting Opioid Misuse
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0433
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Chronic Non Cancer Pain
Keywords: Opioid; Misuse; Community pharmacy; POMI test

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic non cancer pain: Patients with chronic non cancer pain, treated with opioids and having completed the POMi questionnaire

SUMMARY:
Opioid use is increasing in Western countries and is associated with harms as hospitalization, addiction and deaths(1). Community pharmacists interact frequently with patients, giving them the opportunity to identify and prevent the risk of prescribed opioid misuse. The purpose of this study was therefore to assess the risk of prescribed opioids misuse in ambulatory patients with chronic non-cancer pain (CNCP) seen in community pharmacies.

Method: A questionnaire (including the Prescription Opioid Misuse POMI(2)) have been proposed to patients with opioid prescription by pharmacy students, in 86 pharmacies of Occitanie-Est, in April 2019. Eligible patients were adults with CNCP that consented to participate.

A total of 414 patients (62.4% women, mean age 58 ± 16.00) have been included. The main pains were spinal (37.3%) and osteoarticular (33.1%). The median visual analog scale (VAS) was 7 [IQR25-75: 5-8]. The prescribed opioids are mainly weak opioids (73.2%): paracetamol/tramadol (35%), paracetamol/codeine (17.4%), paracetamol/opium (16.8%). Strong opioids (32.6%) were oxycodone (11.95%), fentanyl (9%), and morphine (9%). The median morphine milligram equivalent (MME) was 40 mg/day [IQR25-75: 20-80].

POMI score was superior to 2/6 in 45.4% and superior to 4 in 16%. The main positive question were feel high (40.3%), take the opioid more often (39.3%), take more medication (36.6), and need to early renew opioid medication earlier (30.8%).

Patients with POMI score > 4 were younger (49 years versus 55.9; p<0.01), more urban (78.1% versus 69.2%; p=0.03), had higher VAS (7.3 versus 6.2; p<0.01), received higher median MME (112 mg versus 64.9 mg; p<0.01), and consumed more strong opioid (45.3% versus 27.3%; p=0.04).

ELIGIBILITY:
Inclusion criteria:

* -Collection of the questionnaire in a community pharmacy of the area of investigation East-Occitania)
* Patient over 18 years of age
* Suffering from pain (CNCP) (> 3 months old)
* Treated with weak or strong opioids

Exclusion criteria:

* Collection of the questionnaire in a community pharmacy outside Eastern Occitania
* Patient under 18 years of age
* Suffering from acute pain (< 3 months old) or cancerous pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic non cancer pain
Sampling Method: Non-Probability Sample
Enrollment: 414 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Patients with POMI test "Prescribed Opioid Misuse Index"> 2 | 1 day
  Patients with POMI test > 2 A score >2, may be associated with a risk of misuse of opioid medication. It is recommended to discuss this with the physician

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Peyrière, PH, Principal Investigator — UH Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC